CLINICAL TRIAL: NCT00398320
Title: A Phase II Study of Capecitabine, Oxaliplatin and Bevacizumab for Metastatic or Unresectable Neuroendocrine Tumors
Brief Title: Phase II Capecitabine, Oxaliplatin & Bevacizumab for Metastatic / Unresectable Neuroendocrine Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pamela L. Kunz (Other)
Responsible Party: Sponsor-Investigator, Pamela L. Kunz, Assistant Professor of Medicine, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-06233; 97273; NET0002 (Other: OnCore); NCT00398320; END0002 (formerly) (Other: OnCore)
Record Dates: First submitted 2006-10-31; First posted 2006-11-10 (Estimated); Results first posted 2013-12-10 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-01

CONDITIONS: Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Capecitabine; Oxaliplatin; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bevacizumab (Avastin), Oxaliplatin (Eloxatin) (Experimental)
  Interventions: Drug: Capecitabine; Drug: Oxaliplatin; Drug: Bevacizumab

INTERVENTIONS:
Drug: Capecitabine — 850 mg/m2 by mouth twice a day for days 1-14 oa a 21 day cycle
Drug: Oxaliplatin — 130 mg/m2 intravenously on day 1 of a 21 day cycle
Drug: Bevacizumab — 7.5mg/kg Intravenous on day 1 of a 21 day cycle

SUMMARY:
Given the lack of other viable treatment options for metastatic neuroendocrine tumors, contrasted with our positive anecdotal experience, and the relative tolerability of the treatment regimen for colorectal cancer patients, we propose a single-institution phase II trial investigating the efficacy of capecitabine, oxaliplatin and bevacizumab for patients with metastatic neuroendocrine tumors.

DETAILED DESCRIPTION:
PRIMARY

1. Determine an estimation of median time to progression (TTP) for patients treated with bevacizumab in combination with capecitabine and oxaliplatin
2. Assess the toxicities associated with this regimen

SECONDARY

1. Determine objective response rate (RR) for patients treated with this regimen
2. Conduct exploratory analyses of efficacy according to degree of tumor differentiation and primary location
3. Determine utility of biochemical markers as a surrogate endpoint for tumor response

ELIGIBILITY:
Inclusion Criteria: Subjects must be treated at Stanford University Medical Center for the entire length of study participation.

* Patients must have histologically or cytologically confirmed neuroendocrine tumor, including both well-differentiated tumors (carcinoid) or moderately to poorly differentiated tumors. Patients must be deemed unresectable due to involvement of critical vasculature, adjacent organ invasion, or presence of metastasis.
* Patients with prior surgical resection who develop radiological or clinical evidence of metastatic cancer do not require separate histological or cytological confirmation of metastatic disease unless an interval of > 5 years has elapsed between the primary surgery and the development of metastatic disease. Clinicians should consider biopsy of lesions to establish diagnosis of metastatic disease if there is substantial clinical ambiguity regarding the nature or source of apparent metastases.
* Prior chemotherapy will be permitted, although the patient may not have had prior oxaliplatin.
* Patients must have a primary or metastatic lesion measurable in at least one dimension by Modified RECIST criteria (see Section 4.2) within 4 weeks prior to entry of study
* Patients must have Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* Patients must be ≥ 18 years of age
* Laboratory values ≤ 2 weeks prior to randomization:

  * Absolute Neutrophil Count (ANC) >=1500/mm3
  * Platelets (PLT) ≥ 100,000/mm3
  * Hemoglobin (Hgb) ≥ 9 g/dL
  * Serum creatinine ≤ 1.5 x upper limit of normal (ULN)
  * Serum bilirubin ≤ 1.5 x ULN (≤ 3.0 x ULN if liver metastases present)
  * Aspartate aminotransferase (AST/SGOT), alanine aminotransferase (ALT/SGPT), and alkaline phosphatase ≤ 3.0 x ULN (≤ 5.0 x ULN if liver metastases present). Note: Endoscopic retrograde cholangiopancreatogram (ERCP) or percutaneous stenting may be used to normalize the liver function tests.
* Life expectancy ≥ 12 weeks
* Ability to give written informed consent according to local guidelines

Exclusion Criteria:- Disease-Specific Exclusions

1. Prior oxaliplatin for any reason.
2. Prior full field radiotherapy ≤ 4 weeks or limited field radiotherapy ≤ 2 weeks prior to enrollment. Patients must have recovered from all therapy-related toxicities. The site of previous radiotherapy should have evidence of progressive disease if this is the only site of disease.
3. Prior biologic or immunotherapy ≤ 2 weeks prior to registration. Patients must have recovered from all therapy-related toxicities
4. Prior therapy with anti-vascular endothelial growth factor (VEGF) agents
5. If history of other primary cancer, subject will be eligible only if she or he has:

   * Curatively resected non-melanomatous skin cancer
   * Curatively treated cervical carcinoma in situ
   * Other primary solid tumor curatively treated with no known active disease present and no treatment administered for the last 3 years
6. Concurrent use of other investigational agents and patients who have received investigational drugs ≤ 4 weeks prior to enrollment.

   * General Medical Exclusions

1. Subjects known to have chronic or active hepatitis B or C infection 2. History of any medical or psychiatric condition or laboratory abnormality that in the opinion of the investigator may increase the risks associated with study participation or study drug administration or may interfere with the conduct of the study or interpretation of study results 3. Male subject who is not willing to use adequate contraception upon enrollment into this study and for 6 months following the last dose of second-line treatment 4. Female subject (of childbearing potential, post-menopausal for less than 6 months, not surgically sterilized, or not abstinent) who is not willing to use an oral, patch or implanted contraceptive, double-barrier birth control, or an intrauterine device (IUD) during the course of the study and for 6 months following the last dose of second-line treatment 5. Female subject who is breast-feeding or who has positive serum pregnancy test 72 hours prior to randomization 6. Pleural effusion or ascites that causes respiratory compromise (≥ CTCAE grade 2 dyspnea) 7. Any of the following concurrent severe and/or uncontrolled medical conditions within 24 weeks of enrollment which could compromise participation in the study:

* Unstable angina pectoris
* Symptomatic congestive heart failure
* Myocardial infarction ≤ 6 months prior to registration and/or randomization
* Serious uncontrolled cardiac arrhythmia
* Uncontrolled diabetes
* Active or uncontrolled infection
* Interstitial pneumonia or extensive and symptomatic interstitial fibrosis of the lung
* Chronic renal disease
* Acute or chronic liver disease (eg, hepatitis, cirrhosis) 8. Patients unwilling to or unable to comply with the protocol 9. Life expectancy of less than 12 weeks 10. Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study other than a Genentech-sponsored bevacizumab cancer study

  * Bevacizumab-Specific Exclusions

    1. Inadequately controlled hypertension (defined as systolic blood pressure > 150 and/or diastolic blood pressure > 100 mmHg on antihypertensive medications)
    2. Any prior history of hypertensive crisis or hypertensive encephalopathy
    3. New York Heart Association (NYHA) Grade II or greater congestive heart failure (see Appendix E)
    4. History of myocardial infarction or unstable angina within 6 months prior to study enrollment
    5. History of stroke or transient ischemic attack within 6 months prior to study enrollment
    6. Known central nervous system (CNS) disease
    7. Significant vascular disease (eg, aortic aneurysm, aortic dissection)
    8. Symptomatic peripheral vascular disease
    9. Evidence of bleeding diathesis or coagulopathy
    10. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study enrollment or anticipation of need for major surgical procedure during the course of the study
    11. Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to study enrollment
    12. History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to study enrollment
    13. Serious, non-healing wound, ulcer, or bone fracture
    14. Urine protein ≥ 2+ on urinalysis dipstick and ≥ 1.0 gram on 24-hour urine collection
    15. Known hypersensitivity to any component of bevacizumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-11; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela L Kunz, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled at one site in the US over a three-year period.
Groups:
- Capecitabine / Oxaliplatin / Bevacizumab: Oxaliplatin: 130 mg/m2 intravenously on day 1 of a 21-day cycle
  Capecitabine: 850 mg/m2 by mouth twice a day for days 1 to 14 on a 21-day cycle
  Bevacizumab: 7.5mg/kg intravenously on day 1 of a 21-day cycle
  Adverse events (AEs) reported are related and grade 3 or higher per CTCAE version 3.
Period: Overall Study
Arm/Group | Capecitabine / Oxaliplatin / Bevacizumab
Started | 40
Completed | 34
Not Completed | 6
Not completed — Death | 1
Not completed — Adverse Event | 4
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Groups:
- Capecitabine / Oxaliplatin / Bevacizumab: Oxaliplatin: 130 mg/m2 intravenously on day 1 of a 21-day cycle
  Capecitabine: 850 mg/m2 by mouth twice a day for days 1 to 14 on a 21-day cycle
  Bevacizumab: 7.5mg/kg intravenously on day 1 of a 21-day cycle
  AEs reported are related and grade 3 or higher per CTCAE version 3.
Arm/Group | Capecitabine / Oxaliplatin / Bevacizumab
Number analyzed (Participants) | 40
Age, Continuous [Median (Full Range); unit: years] | 55 [32 to 76]
Gender [Count of Participants; unit: Participants]
  Female | 18
  Male | 22
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: 12-month Progression Free Survival (PFS)
Description: Percentage of participants with 12-month progression-free survival (PFS) was assessed. PFS is defined as the time from enrollment until documented disease progression or death (whichever occurred first). RECIST criteria (version 1). Complete response (CR) defined as disappearance of all target lesions. Partial Response (PR) defined as ≥ 30% decrease of SLD. Progressive disease (PD) defined as ≥ 20% increase in Sum Longest Diameters (SLD). Stable Disease (SD) defined as being between 20% increase and < 30% decrease in SLD.
Time Frame: PFS assessed every 3 months through 12 months
Measure: Number; unit: percentage of participants w/ 12 mo PFS
Arm/Group | Capecitabine / Oxaliplatin / Bevacizumab
Number analyzed (Participants) | 40
percentage of participants w/ 12 mo PFS | 64.7

2. Primary Outcome: Number of Patients Who Experienced Treatment-related Grade 3 or Higher Adverse Events by CTCAE Version 3.0
Description: Participants were monitored every 3 weeks while on study. Toxicity and attributions were as per CTCAE version 3.0 guidelines. Analysis population below is patient who experienced related Grade 3 or higher AE; denominator is 40 total patients enrolled.
Time Frame: 30 days after last treatment
Measure: Number; unit: participants
Arm/Group | Capecitabine / Oxaliplatin / Bevacizumab
Number analyzed (Participants) | 40
participants | 28

3. Secondary Outcome: Response Rates
Description: Response rate is defined as percent of patients with complete response (CR) and partial response (PR) as their best response as defined by RECIST criteria (version 1). Complete response (CR) is defined as disappearance of all target lesions. Partial Response (PR) is defined as ≥ 30 decrease in the sum of longest diameters of target lesions (SLD). Overall response (OR) = CR + PR.
Time Frame: Response rates by RECIST criteria assessed every 3 months while on treatment
Measure: Number; unit: percentage of participants
Arm/Group | Capecitabine / Oxaliplatin / Bevacizumab
Number analyzed (Participants) | 40
percentage of participants | 17.5

4. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as time from enrollment until death from any cause.
Time Frame: Continuous
Measure: Median (Full Range); unit: months
Arm/Group | Capecitabine / Oxaliplatin / Bevacizumab
Number analyzed (Participants) | 40
months | 42.2 [0.6 to 60.8]

5. Secondary Outcome: Biochemical Markers
Time Frame: Assessed every 3 weeks while on treatment
Population: 18 of 40 patients had elevated baseline hormone markers, including Chromogranin A, Gastrin, Glucagon, Pancreatic Polypeptide, vasoactive intestinal peptide (VIP), Urine 5HIAA
Measure: Number; unit: participants
Arm/Group | Capecitabine / Oxaliplatin / Bevacizumab
Number analyzed (Participants) | 18
participants
  25 to 49% reduction in 1 or more hormones | 6
  ≥ 50% reduction in 1 or more hormones | 12

ADVERSE EVENTS:
Time Frame: AEs were collected approximately every 3 weeks when patients were seen by treating MD while they were on active treatment.
Description: If a subject experiences more than one of a given AE, the subject is counted only once for that AE.
Arm/Group | Capecitabine / Oxaliplatin / Bevacizumab
Serious Adverse Events (participants affected / at risk) | 14/40
Other Adverse Events (participants affected / at risk) | 20/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Capecitabine / Oxaliplatin / Bevacizumab (N=40)
Thrombosis/Embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Syncope (Nervous system disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3)
Death (General disorders) | 1 (1)
Confusion (Nervous system disorders) | 1 (1)
Wound dehiscence (Surgical and medical procedures) | 1 (1)
Right tongue numbness/deviation (Nervous system disorders) | 1 (1)
Weight loss (General disorders) | 1 (1)
Anorexia (General disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 1 (1)
Hemorrhage, GI (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Capecitabine / Oxaliplatin / Bevacizumab (N=40)
Tinnitus (Ear and labyrinth disorders) | 1
Low hemoglobin (Blood and lymphatic system disorders) | 2
Low leukocytes (Blood and lymphatic system disorders) | 1
Low neutrophils (Blood and lymphatic system disorders) | 2
Hypertension (Cardiac disorders) | 5
Hand foot skin reaction (Skin and subcutaneous tissue disorders) | 4
Dehydration (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 8
Nausea (Gastrointestinal disorders) | 1
Bowel obstruction (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Hemorrhage, GI Upper (Gastrointestinal disorders) | 2
Elevated Alk Phos (Metabolism and nutrition disorders) | 1
Hyperbilirubinemia (Metabolism and nutrition disorders) | 1
Proteinuria (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Sensory neuropathy (Nervous system disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 2
Headache (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No